CLINICAL TRIAL: NCT02395939
Title: Randomised Controlled Trial Comparing the Diagnostic Yield of Radial Endo-Bronchial Ultra-Sound (R-EBUS) Guided Cryo-biopsy Vs. CT-guided Transthoracic Biopsy in Patients With Parenchymal Lung Lesion, Suspected of Lung Cancer (CT-CROP)
Brief Title: Comparing Diagnostic Yield Between R-EBUS Guided Cryo Biopsy Vs. CT Guided Biopsy for PPL
Acronym: CT-CROP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Middlemore Hospital, New Zealand (Other)
Responsible Party: Principal Investigator, Samantha Herath, Respiratory Physician, Intervetional bronchoscopist, Middlemore Hospital, New Zealand
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CT-CROP
Record Dates: First submitted 2015-03-08; First posted 2015-03-24 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Lung Cancer
Keywords: Cryobiopsy; Radial EBUS; Guide Sheath; Peripheral pulmonary lesions
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CT guided core biopsy (Active Comparator): In patients allocated to this arm a CT guided core biopsy will be performed
  Interventions: Procedure: CT guided core biopsy
- Cryo-biopsy via Radial EBUS navigation (Active Comparator): If the patient is randomised to this arm, the lesion will be located via R-EBUS.
  Each patient will have 3 cryo biopsies and 3 forceps biopsies. The order of the cryo biopsy and forcep biopsy will be randomly allocated at the time of initial randomisation.
  Interventions: Procedure: Cryo-biopsy via Radial EBUS navigation

INTERVENTIONS:
Procedure: CT guided core biopsy — CT guided biopsy will be performed by a trained interventional radiologist using core biopsy.
  Arms: CT guided core biopsy
Procedure: Cryo-biopsy via Radial EBUS navigation — Cryo-biopsy will be performed via R-EBUS guidance. Cryo biopsy probe will be applied for 4 seconds for each biopsy and a minimum of 3 biopsies will be performed . Each patient will also have 3 forceps biopsies. The order of forceps biopsy or cryo biopsy will be randomly allocated.
  Arms: Cryo-biopsy via Radial EBUS navigation

SUMMARY:
Obtaining a tissue sample to diagnose a PPL suspected of cancerous origin is of utmost importance. The current gold standard; Transthoracic CT guided needle biopsy approach with a success rate of >90% comes at the expense of an increased side effect profile.

Given that most lung cancers originate in the bronchus, hence named "bronchogenic carcinoma", it would be rational to think that endobronchial route should provide the best route of sampling with the least amount of side effects. Radial EBUS has become popular during the last decade as an endobronchial modality in diagnosing PPL with minimal side effects. However, the yield is still not satisfactory in comparison to CT guided biopsy with only 73% success rate in a meta-analysis. There is also with wide variation in different centres.

Use of a new biopsy method called cryo-biopsy using the R-EBUS guide sheath may bridge the gap and increase the diagnostic yield of PPL.

Cryo biopsy had been proven to give larger sample sizes and reduced crush artefact compared to the conventional radial EBUS biopsies.

However, there have been no head to head trials comparing Cryo-probe biopsy vs. the gold standard: CT guided biopsy.

Cryo-biopsy has very favourable side effect profile without any pneumothorax occurrence. If the yield were to be non-inferior to CT guided biopsy this would certainly be the preferred choice of biopsy for PPL in the future.

Methodology All patients with a PPL requiring a diagnostic biopsy will be eligible for recruitment to the trial. The recruited patients will be randomly allocated to either CT guided core biopsy or radial EBUS guided cryobiopsy.

Study design Multi centre intervetional,randomised control trial.

Study population:

Patients diagnosed with a PPL that requires a biopsy.

If the patient is randomised to the cryo biopsy arm:

The procedure will be done under the usual guidelines and practice of the centre as for a flexible bronchoscopy procedure.

Once flexible bronchoscopy is introduced the pre-determined desired segment, the R-EBUS is inserted covered by the GS.

Once the R EBUS locates the lesion, the GS is left in situ and the USS probe is retracted.

The cryoprobe is then inserted through the GS to the desired location. Flexible Cryoprobe (outer diameter 1.9mm) will be applied for 4 seconds for each biopsy. The cryogen gas used will be Co2.

The probe will be retracted together with the GS and the bronchoscope en masse after each biopsy. A minimum of 1 and maximum of 3 samples will be taken.

A CXR is taken within 1 hour post procedure to access for pneumothorax. Adverse events during the procedure will be recorded. If a chest tube placement, other investigations due to side effects or overnight hospital stay were to be required; all costs will be calculated retrospectively. Minor bleeding will not be considered an additional cost as this occurs with routine bronchoscopy.

If the patient is randomised to the CT biopsy arm:

A CT guided core biopsy will be performed as per usual practice of that centre. 2-6 passes will be performed for each PPL.

A CXR 1hour post procedure will be performed to assess for pneumothorax or procedure related bleeding.

If a chest tube placement, other investigations due to side effects or overnight hospital stay were to be required all costs will be calculated retrospectively.

At the pathology:

All samples will be assessed for the size of the sample and the suitability for molecular testing. An independent pathologist will assess samples.

Economic analysis:

For both procedures: Both direct and indirect costs will be calculated. The main aim of cost analysis is to calculate the cost of side effect management in each arm to determine the most cost-effective method of sampling a PPL.

DETAILED DESCRIPTION:
Obtaining a tissue sample to diagnose PPL suspected of cancerous origin is of utmost importance. Sampling of PPL can be done either through the chest wall (transthoracic) or through the airways that lead to the PPL (endobronchial).

The current gold slandered is Transthoracic Needle Aspiration (TTNA) approach is done by using CT guided biopsy with a success rate of >90%. However, this success in diagnostic yield comes at the expense of increased side effect profile including a very high risk of pneumothorax (up to 30%). Half of these patients require chest drain insertion.

Given that most lung cancers originate in the bronchus, hence named "bronchogenic carcinoma", it would be rational to think that endobronchial route should provide the best way of sampling with least amount of side effects. However, the yield is still not satisfactory and has a wide confidence interval.

When diagnosing a PPL endobronchially, accurate visualisation of the lesion is the main issue. To overcome this issue various navigation methods have been used to accurately locate the PPL to improve the diagnostic yield.

The use of Radial Endo Bronchial USS (R-EBUS) is one such navigational modality. The conventional R-EBUS guided biopsies are carried out using cytology brushes and forceps biopsy. These methods had been extremely safe with <1% pneumothorax rate however, the diagnostic yield in a meta-analysis of 14 studies is only 73%.

Use of a new biopsy method called cryo-biopsy may bridge the gap and increase the diagnostic yield of PPL.

Cryotherapy is the use of a compressed gas released at a high flow that rapidly expands and creates very low temperatures up to -89C. These very low temperatures then cause tissue to get stuck to the end of the cryo-probe. Due to the rapid cooling the microvasculature around the biopsy site go into vasospasm and reduces bleeding despite a large biopsy sample being acquired.

Cryotherapy has been used in the airway since 1968. The ability to use this method while the patient is using high flow oxygen as well as being a cheap equipment to use makes it very affordable and useful equipment in any interventional bronchoscopy unit. Most bronchoscopists will be trained and familiar with cryo biopsy technique.

The cryo-biopsies were compared against forceps biopsies in this study and demonstrated larger sample size and less crush artefact favouring cryo- biopsy use.

The most encouraging results published recently was looking at cryo-biopsy for PPL using R-EBUS guidance, which demonstrated a yield of 74% and the ability to obtain 3 times larger tissue biopsies when compared to traditional forceps biopsies. There were no pneumothorax in this cohort and only minor bleeding was recorded requiring bronchoscopy suction alone and no other intervention recorded.

However, there had been no head to head trials comparing Cryo-probe vs. the gold standard: CT-guided biopsy.

As cryo-biopsy has very favourable side effect profile without any pneumothorax occurrence if the yield were to be non-inferior this would certainly be the preferred choice of biopsy for PPL in the future.

With regards to cost analysis it has been shown that R-EBUS guided biopsy Vs. CT guided biopsy has similar cost profiles for the procedure alone. However the final cost of the procedure depends on the side effects experienced using each procedure, making CT guided biopsy the costlier of the 2 methods.

However, cryo-biopsy and CT guided biopsy had not been compared in an economic analysis before.

Methodology All patients with a PPL requiring a diagnosis will be eligible for the trial.

Prior to the procedure: (Either CT guided biopsy or cryo biopsy)

1. The size of the lesion will be recorded (volume assessment and maximum diameter on the axial scan) from the CT scan prior to procedure. .

If the patient is randomised to the cryo biopsy arm:

1. The bronchoscopist will plan the pathway to the PPL based on the CT scans. The sub segments from which the lesions could be biopsied will be pre-determined and documented. If available, virtual bronchoscopy will be used to confirm this navigational path to the lesion.
2. Maximum time allowed to locate the lesion via R-EBUS would be 20 mins.
3. The procedure will be done under the usual guidelines and practice of the centre as for a flexible bronchoscopy procedure. As this is a multi-centre trial centre variation on the usual practice of bronchoscopy may vary.
4. Some centres may use fluoroscopy, in addition, to localise the lesion. This is also acceptable in the protocol.
5. If an endobronchial lesion is found then the patient is excluded.
6. Once flexible bronchoscopy is introduced the pre-determined desired segment, the R-EBUS is inserted covered by the GS.
7. Once the R EBUS locates the lesion, the GS is left in situ and the USS probe is retracted.
8. The cryo probe is then inserted through the GS to the desired location. Flexible Cryo probe (outer diameter 1.9 mm) will be applied for 4 seconds for each biopsy.
9. The probe will be retracted together with the GS and the bronchoscope en masse after each biopsy.
10. A minimum of 1 and maximum of 3 samples will be taken.
11. A CXR is taken within 1-hour post procedure to access for pneumothorax.
12. Adverse events during the procedure will be recorded as: Minor bleeding (requiring cold saline or adrenalin), moderate bleeding (requiring a bronchial blocker or APC) and a large bleed (requiring blood transfusion, FFP, cardiothoracic support) etc.
13. If a chest tube placement, other investigations due to side effects or overnight hospital stay were to be required all costs will be calculated retrospectively. Minor bleeding will not be considered an additional cost as this occurs with routine bronchoscopy.

If the patient is randomised to the CT biopsy arm:

1. The interventional radiologist will decide on the best position for the patient to stay during the procedure.
2. A core biopsy will be performed as per usual practice of that centre. In CMDHB all CT guided biopsies are performed as core biopsies.
3. The patient will have 2-6 biopsies from the PPL.
4. Patient lies on the side of the biopsy for 1 hour post procedure. Post procedure monitoring will be performed as per usual practice.
5. A CXR 1 hour post procedure will be performed to assess for pneumothorax or procedure related bleeding.
6. If a chest tube placement, other investigations due to side effects or overnight hospital stay were to be required all costs will be calculated retrospectively.

At the pathology:

All samples will be assessed for area of specimen to assess the size. The ability to perform molecular typing will be documented.

An independent pathologist will assess samples

Economic analysis:

For both procedures: Both direct costs (From the hospital records) and indirect cost (by administering a patient questionnaire) will be recorded.

The main aim of cost analysis is to calculate the cost of side effect management in each arm to determine the most cost effective method of sampling a PPL.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged >18 years with a peripheral pulmonary lesion, suspected of lung cancer, requiring a biopsy
* The lesion will be included irrespective of the relationship to the bronchus or ground glass appearance.

Exclusion Criteria:

1. Patients with mediastinal adenopathy amenable to liner EBUS should have this procedure first and enrolled only if it fails to derive a diagnosis.
2. Endobronchial tumour on flexible bronchoscopy
3. Platelet count>150
4. International Normalised Ratio >=1.5
5. Haemoglobin>100
6. Neutrophils >1.0
7. Glomerular Filtration Rate>30
8. Liver Function Test< 2 times upper limit of normal
9. Unable to give consent/intellectually impaired

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield of cryo biopsy Vs. CT guided biopsy as measured by final histological diagnosis | 2 years
  This outcome measures the efficacy of CT guided biopsy (The current Gold standard) against the new biopsy method called cryo-biopsy which has better safety profile from previous pilot studies.

SECONDARY OUTCOMES:
Safety profile as measured by the rate of pneumothorax and bleeding | 2 years
  The CT guided biopsy has good efficacy rates but a high risk of pneumothorax (up to 30%) and pulmonary haemorrhage (4-27%), which requires further management adding to the cost of the intervention. The cryobiopsy method had been proven in pilot studies to have a better safety profile with <1% pneumothorax risk. Hence comparing the side effect profile and if cryo biopsy is far safer alternative would make this the first option for the patient.
Ability to sub type and molecular type the biopsy sample over and above the conventional radial EBUS samples | 2 years
  Cryo biopsy gives a larger sample size and hypothesized to give a better molecular analysis for EGFR mutation and ALK mutation analysis

OTHER OUTCOMES:
Cost analysis between cryo biopsy and CT guided biopsy for PPL | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Herath, MBBS, FRACP, Principal Investigator — Middlemore Hospital, New Zealand
Locations (1):
- Middlemore Hospital,, Auckland, New Zealand

REFERENCES:
- [Result] National Lung Screening Trial Research Team; Aberle DR, Adams AM, Berg CD, Black WC, Clapp JD, Fagerstrom RM, Gareen IF, Gatsonis C, Marcus PM, Sicks JD. Reduced lung-cancer mortality with low-dose computed tomographic screening. N Engl J Med. 2011 Aug 4;365(5):395-409. doi: 10.1056/NEJMoa1102873. Epub 2011 Jun 29. PMID 21714641
- [Result] Prosch H, Stadler A, Schilling M, Burklin S, Eisenhuber E, Schober E, Mostbeck G. CT fluoroscopy-guided vs. multislice CT biopsy mode-guided lung biopsies: accuracy, complications and radiation dose. Eur J Radiol. 2012 May;81(5):1029-33. doi: 10.1016/j.ejrad.2011.01.064. Epub 2011 Jul 12. PMID 21752567
- [Result] Loh SE, Wu DD, Venkatesh SK, Ong CK, Liu E, Seto KY, Gopinathan A, Tan LK. CT-guided thoracic biopsy: evaluating diagnostic yield and complications. Ann Acad Med Singap. 2013 Jun;42(6):285-90. PMID 23842769
- [Result] Montaudon M, Latrabe V, Pariente A, Corneloup O, Begueret H, Laurent F. Factors influencing accuracy of CT-guided percutaneous biopsies of pulmonary lesions. Eur Radiol. 2004 Jul;14(7):1234-40. doi: 10.1007/s00330-004-2250-3. Epub 2004 Feb 13. PMID 14963689
- [Result] Arslan S, Yilmaz A, Bayramgurler B, Uzman O, Nver E, Akkaya E. CT- guided transthoracic fine needle aspiration of pulmonary lesions: accuracy and complications in 294 patients. Med Sci Monit. 2002 Jul;8(7):CR493-7. PMID 12118196
- [Result] Wu CC, Maher MM, Shepard JA. Complications of CT-guided percutaneous needle biopsy of the chest: prevention and management. AJR Am J Roentgenol. 2011 Jun;196(6):W678-82. doi: 10.2214/AJR.10.4659. PMID 21606253
- [Result] Grasso RF, Cazzato RL, Luppi G, D'Agostino F, Schena E, Del Vescovo R, Giurazza F, Faiella E, Beomonte Zobel B. Percutaneous lung biopsies: performance of an optical CT-based navigation system with a low-dose protocol. Eur Radiol. 2013 Nov;23(11):3071-6. doi: 10.1007/s00330-013-2932-9. Epub 2013 Jun 20. PMID 23783784
- [Result] Hsiao SH, Chung CL, Lee CM, Chen WY, Chou YT, Wu ZH, Chen YC, Lin SE. Suitability of computed tomography-guided biopsy specimens for subtyping and genotyping of non-small-cell lung cancer. Clin Lung Cancer. 2013 Nov;14(6):719-25. doi: 10.1016/j.cllc.2013.06.002. Epub 2013 Jul 25. PMID 23891241
- [Result] S H. CT guided lung biospy-FNA or core biospy? Royal Australian New Zealand College of Radiology 2013;2013 Abstract
- [Result] Gasparini S, Ferretti M, Secchi EB, Baldelli S, Zuccatosta L, Gusella P. Integration of transbronchial and percutaneous approach in the diagnosis of peripheral pulmonary nodules or masses. Experience with 1,027 consecutive cases. Chest. 1995 Jul;108(1):131-7. doi: 10.1378/chest.108.1.131. PMID 7606947
- [Result] Baaklini WA, Reinoso MA, Gorin AB, Sharafkaneh A, Manian P. Diagnostic yield of fiberoptic bronchoscopy in evaluating solitary pulmonary nodules. Chest. 2000 Apr;117(4):1049-54. doi: 10.1378/chest.117.4.1049. PMID 10767238
- [Result] Schuhmann M, Bostanci K, Bugalho A, Warth A, Schnabel PA, Herth FJ, Eberhardt R. Endobronchial ultrasound-guided cryobiopsies in peripheral pulmonary lesions: a feasibility study. Eur Respir J. 2014 Jan;43(1):233-9. doi: 10.1183/09031936.00011313. Epub 2013 Jul 30. PMID 23900983
- [Result] Steinfort DP, Liew D, Irving LB. Radial probe EBUS versus CT-guided needle biopsy for evaluation of peripheral pulmonary lesions: an economic analysis. Eur Respir J. 2013 Mar;41(3):539-47. doi: 10.1183/09031936.00044612. Epub 2012 Jul 26. PMID 22835609
- [Result] Griff S, Ammenwerth W, Schonfeld N, Bauer TT, Mairinger T, Blum TG, Kollmeier J, Gruning W. Morphometrical analysis of transbronchial cryobiopsies. Diagn Pathol. 2011 Jun 16;6:53. doi: 10.1186/1746-1596-6-53. PMID 21679402
- [Result] Hetzel J, Eberhardt R, Herth FJ, Petermann C, Reichle G, Freitag L, Dobbertin I, Franke KJ, Stanzel F, Beyer T, Moller P, Fritz P, Ott G, Schnabel PA, Kastendieck H, Lang W, Morresi-Hauf AT, Szyrach MN, Muche R, Shah PL, Babiak A, Hetzel M. Cryobiopsy increases the diagnostic yield of endobronchial biopsy: a multicentre trial. Eur Respir J. 2012 Mar;39(3):685-90. doi: 10.1183/09031936.00033011. Epub 2011 Aug 18. PMID 21852332